CLINICAL TRIAL: NCT07051304
Title: Evaluation of Patient Preference and Interpretability of Video-Based Pain Expression Scenarios Compared to the Numerical Rating Scale (NRS) in the Postoperative Period: A Prospective Single-Center Pilot Study
Brief Title: Video-Based Versus Numerical Pain Assessment in Postoperative Patients: A Pilot Study
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Engin Ihsan Turan, principal investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: pain assesment with videos
Record Dates: First submitted 2025-06-25; First posted 2025-07-04 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pain Assessment Scales

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: numerical rating scale — The Numerical Rating Scale (NRS) is a standardized, self-reported pain assessment tool in which patients are asked to rate their pain intensity on a scale from 0 to 10.
  0 represents "no pain"
  10 represents "the worst pain imaginable"
Other: Video-Based Pain Expression Scenarios — This novel pain assessment method involves showing postoperative patients a set of pre-recorded video scenarios that visually represent different levels of pain intensity. The videos are 8 seconds long and were created using AI-generated scripts and VEO-3 software. Each scenario corresponds to a specific Numerical Rating Scale (NRS) range (1-2, 3-4, 5-6, 7-8, 9-10) and is portrayed by actors matched to the patient's age group and gender (18-44, 45-65, >65 years; male and female versions available).
  Participants are asked to watch the full video set and select the one that best represents their current postoperative pain experience. This intervention is designed to offer a visual and contextual method of pain expression, particularly beneficial for patients who have difficulty understanding or using abstract numerical scales.

SUMMARY:
The goal of this observational pilot study is to evaluate whether video-based visual scenarios representing different levels of pain are preferred over the traditional Numerical Rating Scale (NRS) by postoperative patients. The study also investigates the clarity and interpretability of both methods and examines the level of agreement between the selected video and the reported NRS score.

DETAILED DESCRIPTION:
This prospective, observational, single-center pilot study evaluates the usability and preference of a novel video-based pain expression method compared to the standard Numerical Rating Scale (NRS) in postoperative adult patients. Videos representing 5 different pain intensities (NRS 1-2, 3-4, 5-6, 7-8, 9-10) were created using AI-assisted scenario generation and VEO-3 video production tools. Each video features age- and sex-matched models (male and female in three age categories: 18-44, 45-65, >65 years) demonstrating realistic, simulated pain expressions.

In the recovery unit, patients aged 18 and above will be shown the video series and asked to:

Select the video that best reflects their current pain

Report their pain using the NRS

Indicate which method (video or NRS) they prefer for expressing pain

Indicate which method they found easier to understand

Collected data will include demographic variables, surgical details, comorbidities, and responses to the pain assessment tools. The study will enroll at least 82 participants based on power analysis.

Data will be anonymized and analyzed using descriptive and inferential statistics including Chi-square, Spearman correlation, and p<0.05 significance level.

The planned sample size was amended prior to the enrollment of the first patient, increasing from 120 to 240 participants. This adjustment was made to ensure sufficient statistical power for planned subgroup analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Undergoing any type of surgery
* Admitted to the postoperative recovery unit (PACU) in stable condition
* Able to understand and respond to questions
* Provide written informed consent (ICF)

Exclusion Criteria:

* Age < 18 years
* Refusal or inability to provide informed consent
* Visual impairment or blindness
* Impaired consciousness or cognitive inability to complete the questionnaire
* History of psychiatric illness
* Planned postoperative ICU admission
* Patients undergoing surgery for intracranial mass
* History of seizure disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult postoperative patients (aged 18 years and older) who are recovering in the recovery room following any type of surgery. Participants must be conscious, cooperative, and capable of evaluating and expressing their pain using both video-based scenarios and the Numerical Rating Scale (NRS). All participants will provide written informed consent prior to participation. The population will include a range of age and gender groups to allow evaluation of method preference across demographic subgroups.
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2025-10-15 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2026-01-04 (Actual)

PRIMARY OUTCOMES:
Patient Preference Between Video-Based and Numerical Rating Scale (NRS) Pain Assessment Methods | Immediately after postoperative evaluation in the recovery unit (within 1 hour after surgery)
  This outcome evaluates which pain assessment method patients prefer after being exposed to both the video-based pain expression scenarios and the traditional NRS scale. Patients will be asked, "Which method did you prefer to express your pain?" and their answers (Video or NRS) will be recorded. The result will be reported as the proportion of participants preferring each method.

SECONDARY OUTCOMES:
Concordance Between Selected Video and Reported NRS Score | Immediately after postoperative evaluation
  Assesses the degree of agreement between the video that the patient selects to represent their pain and the corresponding NRS score they provide.
Perceived Clarity of Pain Assessment Methods | Immediately after postoperative evaluation
  Evaluates which method (Video or NRS) patients found easier to understand. Patients will answer the question: "Which method was easier for you to understand when expressing your pain?" The outcome will be reported as the frequency and percentage distribution of preferences.
Influence of Demographics on Method Preference | Immediately after postoperative evaluation
  This outcome will analyze whether age or sex affects the patient's preference for either the video-based or NRS method. Subgroup analysis will be performed to explore trends in preference across different demographic categories.

CONTACTS AND LOCATIONS:
Overall Officials: Engin ihsan Turan, Specialist, Principal Investigator — Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital
Locations (1):
- Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided